CLINICAL TRIAL: NCT00101075
Title: Phase II Study of Capecitabine and Oxaliplatin (XELOX) in Patients With Locally Advanced, Incurable, Salivary Gland Cancers
Brief Title: Title XELOX FOR SALIVARY GLAND CANCERS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Sanofi-Synthelabo (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-149; P30CA006516 (NIH); SANOFI-DFCI-04149
Record Dates: First submitted 2005-01-07; First posted 2005-01-10 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Head and Neck Cancer
Keywords: high-grade salivary gland mucoepidermoid carcinoma; low-grade salivary gland mucoepidermoid carcinoma; salivary gland acinic cell tumor; salivary gland adenocarcinoma; salivary gland adenoid cystic carcinoma; salivary gland malignant mixed cell type tumor; salivary gland poorly differentiated carcinoma; salivary gland squamous cell carcinoma; recurrent salivary gland cancer; stage III salivary gland cancer; stage IV salivary gland cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Salivary Gland Neoplasms | interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- XELOX (Experimental): * Oxaliplatin 130 mg/m2 day 1 every 3 weeks
  * Capecitabine 1700 mg/m2/day days 1-14 every 3 weeks. -- Patients will be evaluated for response at the end of cycle 2 and at the end of every even cycle thereafter.
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Capecitabine
  Other Names: Xeloda
Drug: Oxaliplatin
  Other Names: Eloxatin

SUMMARY:
The goal of this clinical research study is to find out how effective oxaliplatin and capecitabine are against advanced cancer of the salivary gland. The safety of this treatment as well as how long the cancer responds or stays in a stable state due to the treatment will also be studied.

DETAILED DESCRIPTION:
This is a study of two investigational agents called oxaliplatin and capecitabine.

Investigational agents have not received Food and Drug Administration (FDA) approval for the way they are being used in this study. This means an investigation drug is still under study to determine what a safe dose is, what the side effects are and whether or not it is effective in the disease or condition being studied.

Oxaliplatin and capecitabine are chemotherapy agents that have been approved by the FDA for use in other cancers.

ELIGIBILITY:
Inclusion Criteria

* Histologic diagnosis of any of the following malignancies originating from salivary tissue: adenoid cystic carcinoma, mucoepidermoid carcinoma, acinic cell carcinoma, malignant mixed tumor, polymorphous low grade adenocarcinoma, undifferentiated carcinoma, squamous cell carcinoma, adenocarcinoma.
* Patients must be incurable on the basis of unresectable local or distant disease as determined by the patient's surgeon and not be potentially curable by radiation therapy as determined by a radiation oncologist.
* Patients may have received radiation to any site with the following caveat: the sites used for evaluation for response are either not previously irradiated or they have shown progression of disease post radiation and there has been a time interval of one month since these sites were radiated.
* Patients must have an ECOG performance status of less than 3.
* Patients must have at least uni-dimensionally measurable disease documented within one month of initiation of treatment. Measurement may be by physical exam or radiologically. Attempts should be made to photo document all tumor sites assessed by physical examination with a metric ruler within the photo for measurement confirmation.
* Patients must be willing and able to go through the process of informed consent.
* Patients must have a life expectancy exceeding 3 months.
* Patients must be at least 18 years old.
* Patients must have adequate organ function as defined by the following tests to be performed within 14 days of therapy initiation:

  * Absolute neutrophil count > 1999 cells x 10 6/L
  * Platelet count > 99,999 cells x 10 6/L
  * Hemoglobin >8.5 gm/di or HCT > 25%
  * Serum creatinine < 1.5 x institutional upper limits of normal (ULN) or creatinine clearance measured by 24 hour urine collection as at least 50% of institutional lower limit of normal.
  * Total bilirubin <2 x institutional ULN
  * AST (SGOT) <2 x institutional ULN*

    * * If from documented liver involvement with cancer, may be up to < 5 x institutional ULN Alkaline Phosphatase < 5 x institutional ULN #
    * # If from documented bone or liver involvement with cancer, no upper limit restriction.
* Subjects (male or female) must agree to use effective methods of birth control while on study.
* Subjects should be able to tolerate and swallow tablets or undergo GI tube insertion.

Exclusion Criteria

* Patients must have not received cytotoxic chemotherapy for metastatic salivary gland cancer. Previous immunologic, hormonal, homeopathic, natural, or alternative medicine therapies are acceptable provided treatment ended greater than 28 days prior to protocol therapy. Patients may have received chemotherapy given concomitantly with radiation therapy in an adjuvant setting with curative intent.
* Patients must not receive any form (including radiotherapeutic, immunologic, hormonal,homeopathic, natural, or alternative medicine) of anti-neoplastic therapy other than XELOX while participating in this study.
* Patients must not have a history of any invasive neoplasm within three years of trial entry, excepting curatively treated non-melanoma skin cancer and cervical cancer.
* Pregnant and breast feeding women are not eligible for this study. No pregnancy test is required. Women of childbearing potential must be counseled on the use of effective birth control prior to participation in this study.
* Patients with significant active illness (e.g. congestive heart failure, COPD, uncontrolled diabetes) are not eligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-10; Primary Completion 2007-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Tumor response rate as assessed by RECIST criteria at every 2 courses of treatment | Every 2 Cycles

SECONDARY OUTCOMES:
Progression-free survival as assessed by RECIST criteria at every 2 courses of treatment | Every 2 Cycles
Toxicity as assessed by CTCAE weekly | Weekly
Expression of signal transduction and cell cycle regulatory proteins as assessed by biopsy at baseline and day 3 | Baseline andDay 3

CONTACTS AND LOCATIONS:
Overall Officials: Robert I. Haddad, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No